CLINICAL TRIAL: NCT05416333
Title: A Pilot Study of Azelaic Acid as a Novel Treatment for Central Centrifugal Cicatricial Alopecia
Brief Title: Azelaic Acid as a Novel Treatment for Central Centrifugal Cicatricial Alopecia (CCCA)
Acronym: (CCCA)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00076717
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Central Centrifugal Cicatricial Alopecia
Keywords: hair growth; hair follicle regrowth; hair loss regression
MeSH Terms: interventions — azelaic acid

STUDY DESIGN:
Intervention Model Description: 15 patients for the study will be randomized to one of two groups who consent to participate in a novel treatment with azelaic acid or the control (no additional treatment besides Subject's already prescribed drug)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- azelaic acid treatment (Experimental): Subjects will use the topical formulation once daily on the scalp. The subjects will use the treatment for a total of 6 months.
  Interventions: Drug: azelaic acid
- control (no additional treatment) (Sham Comparator): Subjects will continue to use their current primary provider prescribed topical formulation once daily on the scalp. The subjects will use their treatment for a total of 6 months.
  Interventions: Other: usual medication for CCCA

INTERVENTIONS:
Drug: azelaic acid — Subjects will use the topical formulation once daily on the scalp. The subjects will use the treatment for a total of 6 months
  Other Names: Finacea
  Arms: azelaic acid treatment
Other: usual medication for CCCA — Subjects will continue to use their already prescribed topical formulation once daily on the scalp. The subjects will use their treatment for a total of 6 months
  Arms: control (no additional treatment)

SUMMARY:
The purpose of this pilot study is to determine if azelaic acid shows potential to be an effective treatment for Central Centrifugal Cicatricial Alopecia (CCCA). In this study, the aim is to compare azelaic acid vs placebo since azelaic acid may increase anti-inflammatory effects that affect the hair growth cycle.

DETAILED DESCRIPTION:
The management of Central Centrifugal Cicatricial Alopecia (CCCA) is challenging due to limited current treatments and a lack of randomized controlled trials. Management focuses on behavioral and styling modifications, in addition to symptomatic relief. Any potentially damaging hair care practices such as chemical relaxers, heat application to the scalp, and the use of hardening gels and sprays are discouraged. Many commonly used therapies are anti-inflammatory in nature, including intralesional steroids, topical steroids, oral antibiotics and increased frequency of hair washing with antidandruff shampoos. These treatments not only lead to improvement in pruritus and tenderness, but in some cases result in increased hair density. Currently, comparison studies of different treatments for CCCA subjects is limited. The aim is to determine if there is an advantage in using one particular anti-inflammatory therapy over another for relieving symptoms and promoting hair follicle regrowth.

ELIGIBILITY:
Inclusion Criteria:

* women eighteen years of age or older
* biopsy-proven and /or clinical diagnosis of CCCA Stage II-IV
* on stable treatment without changes for at least three months
* recruited from outpatient dermatology clinics at the Wake Forest Baptist Health Department of Dermatology

Exclusion Criteria:

* males

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males are excluded from this study since the prevalence of CCCA in males is so significantly low that it is difficult to find cases in a clinical setting
Enrollment: 15 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Amount of hair loss regression | Baseline
  measured by standardized photos and dermatoscope photos
Amount of hair loss regression | Month 2
  measured by standardized photos and dermatoscope photos
Amount of hair loss regression | Month 4
  measured by standardized photos and dermatoscope photos
Amount of hair loss regression | Month 6
  measured by standardized photos and dermatoscope photos

SECONDARY OUTCOMES:
Amount of hair regrowth | Months 2, 4, and 6
  measured by standardized photos and dermatoscope photos
Amount of alleviation of signs and symptoms of disease | Months 2, 4, and 6
  Higher scores means worse symptoms and signs of disease - Clinical signs and symptoms of CCCA will be documented by administering a standardized questionnaire to all subjects. Subjects will complete the standardized questionnaire regarding symptoms of their hair loss at the start of the enrollment and every 2 months until the study is completed.
Dermatology Life Quality Index (DLQI) | Baseline and Month 6
  Scores of "not at all" to "very much"

CONTACTS AND LOCATIONS:
Overall Officials: Amy J McMichael, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Scieces, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No